CLINICAL TRIAL: NCT04842838
Title: Comparative Clinical Study of Drug-coating Balloon Strategy and Drug-eluting Stent Strategy in the Treatment of True Bifurcation Coronary Artery Disease
Brief Title: Comparative Clinical Study of Drug-coating Balloon Strategy and Drug-eluting Stent Strategy
Acronym: Kissing-DCB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAW-PMS-R01-01
Record Dates: First submitted 2021-04-02; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB strategy (Experimental)
  Interventions: Device: paclitaxel DCB
- DES strategy (Active Comparator)
  Interventions: Device: DES

INTERVENTIONS:
Device: paclitaxel DCB — Drug-coated balloon is a new kind of coronary interventional device. The balloon coated with anti-cell proliferation drugs (paclitaxel, etc.) is sent to the stenosis site. The balloon is closely adhered to the vascular wall during the expansion, and the drug is rapidly and evenly coated on the disaffected vessels.In recent years, DCB has gradually become an alternative for the treatment of in-stent restenosis (ISR), small vessel disease (SVD) and bifurcation disease.
  Arms: DCB strategy
Device: DES — Provisional T technique is the preferred method for the treatment of bifurcation lesions with the existing stent.According to the 2018 European Guidelines on revascularization and the consensus group of the European Bifurcation Club (EBC), Provisional T technique is still the first choice for the treatment of Bifurcation, despite the problems related to side branches.
  Arms: DES strategy

SUMMARY:
The trial aims to evaluate the long-term clinical outcome of the DCB-only technique is non-inferior to the provisional T stenting with DES in the patients who have 'true' bifurcation lesions.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old;
2. Evidence of myocardial ischemia and indications of PCI, stable or unstable angina pectoris, or old myocardial infarction;
3. Primary and bifurcated coronary artery lesions (Medina classification 1,1,1 or 1,0,1 or 0,1,1);
4. Visual angiography of the main branch reference vessel diameter ≥2.5mm, and ≤4.0mm;Branch reference vessel diameter ≥2.0mm;
5. Diameter stenosis of main and branch lesions ≥ 70%, and diameter stenosis of branch lesions ≥ 50%;
6. Visual examination of residual stenosis of main branch lesions after pre-dilation ≤ 30% without vascular dissection or dissection with NHLBI classification A, B, C type.
7. If 2 bifurcation lesions meet the inclusion requirements, only 1 lesion can be included in the study, and the other lesion can be treated or not treated as a non-target lesion.

Exclusion Criteria:

1. Main branch or branching target lesions require treatment with more than one device (DES or DCB);
2. There is more than 1 non-target lesion requiring intervention on the target blood vessel;
3. The distance between non-target lesion and target lesion is less than 10 mm;
4. Main and branch lesions > 26 mm or branch lesions length BBB> mm;
5. Left main lesion and its bifurcation lesion;
6. Intra-stent restenosis or severe calcification;
7. ST-segment elevation or non-ST-segment elevation myocardial infarction 7 days before surgery;
8. Severe heart failure (NYHA-IV or left ventricular ejection fraction <35%);
9. Cardiogenic shock;
10. known to have renal failure (EGFR <30ml/min/1.73m2);
11. Pregnant or lactating women, or women of reproductive age who had family planning or were unable to take adequate contraceptive measures during the study period;
12. Any known allergic reactions or contraindications to the drug and coating or scaffold metal required for DCB in the study;
13. Other DES or DCB treatment contraindications;
14. Failing to sign an informed consent or having an expected life of less than 12 months;
15. Other researchers consider it inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Target lesion failure (TLF) | 12 months
  Target lesion failure, defined as cardiac death, clinically driven target vessel myocardial infarction and target lesion revascularization.
Number of Participants with net adverse clinical cardiovascular events (NACCE) | 12 months
  Net adverse clinical cardiovascular events, defined as cardiac death, clinically driven target vessel myocardial infarction, target lesion revascularization and major bleeding (BARC type 2, 3, 5 bleeding)

SECONDARY OUTCOMES:
Technical success rate | 1-2 days
  According to CAG, the residual stenosis of the main branch is less than 30% and the residual stenosis of the side branch is less than 50%. The blood flow is of TIMI III as well
Number of Participants with Target lesion failure (TLF) | 1/6/24/36 month
  Target lesion failure, defined as cardiac death, clinically driven target vessel myocardial infarction and target lesion revascularization
Number of Participants with Target lesion revascularization (TLR) | 1/6/12/24/36 month
  Target lesion revascularization, defined as clinically indicated percutaneous or surgical revascularization of the index lesion during follow-up, like using stent, balloon, coronary atherectomy, or CABG
Number of Participants with Target vessel revascularization (TVR) | 1/6/12/24/36 month
  Target vessel revascularization, defined as clinically indicated percutaneous or surgical revascularization of the target vessel during follow-up, like using stent, balloon, coronary atherectomy, or CABG
Clinical procedure time | during the procedure
  The used time in the clinical procedure
DAPT using time | 1/6/12/24/36 month
  The using time of DAPT
Number of Participants with Bleeding events（BARC2, 3, and 5） | 1/6/12/24/36 month
  Definite, probable, or possible thrombus in the device defined by ARC: Acute thrombus, subacute thrombus, late thrombus, and very late thrombus
Number of Participants with ARC defines stent thrombosis | 1/6/12/24/36 month
  The identification and possibility of stent thrombosis were included in the time ranges of acute, subacute, late, and late

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China